CLINICAL TRIAL: NCT02356796
Title: Chronic Pelvic Pain in Women - Conservative Multidisciplinary Group Treatment Compared to Standard Conservative Treatment. A Randomised Controlled Trial.
Brief Title: Chronic Pelvic Pain in Women - Conservative Group Treatment Compared to Standard Conservative Treatment.
Acronym: CPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of North Norway (Other)
Collaborators: The Royal Norwegian Ministry of Health (Other); Norwegian Fund for Postgraduate Training in Physiotherapy (Other); University of Tromso (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014/1398 (REK)
Record Dates: First submitted 2015-02-02; First posted 2015-02-05 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2018-05

CONDITIONS: Pelvis Pain Chronic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Multidisciplinary group treatment (Experimental): Multidisciplinary group intervention at the University Hospital of North Norway. The group intervention is led by physiotherapists, with contributions from a gynecologist, nutritionist and a peer patient. The treatment consists of active exercises and theory lessons. The focus is to enhance the participants body awareness and to recognize the integration of mental and physical processes. The aim is to create change in patterns that influence the participants health negatively.
  The treatment lasts one year. The first meeting has a duration of 10 days, then follow-up after 3, 6 and 12 months.
  Interventions: Other: Multidisciplinary group treatment
- Standard physiotherapy treatment (Active Comparator): Standard treatment in primary or secondary health care physiotherapy. Patients are referred to a physiotherapist with appropriate training/competence, as close to their home as possible.
  Interventions: Other: Standard physiotherapy treatment

INTERVENTIONS:
Other: Multidisciplinary group treatment — Multidisciplinary group intervention at the University Hospital of North Norway. The group intervention is led by physiotherapists, with contributions from a gynecologist, nutritionist and a peer patient. The treatment consists of active exercises and theory lessons. The focus is to enhance the participants body awareness and to recognize the integration of mental and physical processes. The aim is to create change in patterns that influence the participants health negatively.
  The treatment lasts one year. The first meeting has a duration of 10 days, then follow-up after 3, 6 and 12 months.
  Arms: Multidisciplinary group treatment
Other: Standard physiotherapy treatment — Standard treatment in primary or secondary health care physiotherapy. Patients are referred to a physiotherapist with appropriate training/competence, as close to their home as possible.
  Arms: Standard physiotherapy treatment

SUMMARY:
The purpose of this study is to evaluate the effect of a multidisciplinary group based treatment compared to standard physiotherapy for women with chronic pelvic pain (CPP). The hypothesis is that multidisciplinary group based treatment is more effective than standard physiotherapy for women with CPP. The participants will be randomized to one of two treatment arms, and the treatment effect will be evaluated 12 months after start of intervention.

DETAILED DESCRIPTION:
Background: Chronic pelvic pain (CPP) is a common source of pain and reduced quality of life among women throughout the world. CPP is a complex condition, and the understanding of both etiology and effective treatment is limited. The newest/latest clinical guidelines recommend a holistic and multidisciplinary treatment approach to this condition.

In accordance with the guidelines a multidisciplinary group based treatment for women with CPP has been started at the University Hospital of North Norway. The treatment is offered to patients who are considered to benefit from conservative treatment approach.

Method: To investigate the effect of a group based treatment compared to standard conservative treatment by physiotherapists in primary or secondary health care, a randomized controlled trial will be conducted.

Patients who are found eligible and consent to participate in the trial, will be randomized to one of the two treatment options. Data will be registered at baseline, 3, 6 and 12 months after start of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Chronic pelvic pain lasting minimum 6 months
* Motivated for group intervention

Exclusion Criteria:

* Pelvic pathology that needs medical treatment other than conservative
* Pregnancy, or labour last 12 months.
* Abdominal or pelvic surgery the last 6 months
* Botox injections in pelvic areas last 4 months.
* Drug addiction or using large dozes of analgesics
* Serious psychiatric diagnosis. Consent capability is necessary.
* Not speaking/writing Norwegian language
* Previously treated by physiotherapist involved in the group intervention in this project

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2015-02; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Changes in pelvic pain | From baseline to 3, 6 and 12 months after start of intervention.
  Self reported pelvic pain the last 7 days. The worst, the least and the mean pain are recorded. Each item is scored 0-10 (0=no pain, 10 = pain as bad as can be).

SECONDARY OUTCOMES:
Changes in subjective health complaints | From baseline to 3, 6 and 12 months after start of intervention
  Self reported health complaints last 30 days, using a standardized questionnaire.
Changes in fear of movement, | From baseline to 12 months after start of intervention
  Measured with Tampa Scale of Kinesiophobia, a self-completed questionnaire.
Changes in sexual function concerning pain during intercourse | From baseline to 12 months after start of intervention
  Questionnaire recording sexual desire, orgasm problems and pain during intercourse. Each item is scored "all the time", "almost all the time", "often", "rarely" or "never".
Changes in general health condition | From baseline to 3, 6 and 12 months after start of intervention
  EQ-5D questionnaire recording mobility, self-care, usual activities, pain/discomfort and anxiety/depression.
Changes in fecal incontinence, urinary incontinence (UI), obstructed defecation | From baseline to 12 months
  Measured by the standardized St.Marks score, the ICIQ-UI_SF and the Obstructed Defecation Syndrome Score.
Changes in motor functions: posture, movement, gait, sitting posture, respiration | From baseline to 12 months after start of intervention
  A standardized Mensendieck test is used. Motor functions are recorded and evaluated by a trained physiotherapist.

CONTACTS AND LOCATIONS:
Overall Officials: Paal Oian, Professor MD, Study Chair — University Hospital of North Norway
Locations (1):
- University Hospital of North Norway, Tromsø, Troms, Norway